CLINICAL TRIAL: NCT00002937
Title: A Phase II Randomized Study of Paclitaxel Versus Paclitaxel + PSC833 for Advanced Breast Cancer (Recurring Less Than 6 Months Since Adjuvant or as Second Line for Advanced Disease
Brief Title: Paclitaxel With or Without PSC 833 in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065380; U01CA063265 (NIH); CHNMC-96002; NCI-H97-1137
Record Dates: First submitted 1999-11-01; First posted 2004-09-03 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2010-01

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; valspodar

INTERVENTIONS:
Drug: paclitaxel
Drug: valspodar

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Randomized phase II trial to compare the effectiveness of paclitaxel with or without PSC 833 in treating patients with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the response rate and time to treatment failure of paclitaxel with and without the P-glycoprotein (Pgp) antagonist PSC 833 in advanced breast cancer. II. For each treatment arm, relate paclitaxel AUC (area under curve), and/or time above .05 um/L, to myelosuppression and/or response. III. To obtain preliminary estimates of MDR in this group of patients by measuring MDR1-Pgp immunostaining in pretreatment biopsies in 20 patients and biopsies taken at the time of progression.

OUTLINE: This is a randomized study. Patients are stratified according to three criteria: 1) treatment within 2 years of adjuvant chemotherapy vs. progression on chemotherapy for advanced disease 2) measurable vs. evaluable disease 3) institution. Patients receive paclitaxel alone or paclitaxel plus PSC 833. In the first arm, paclitaxel alone is administered by continuous infusion over 3 hours once every 3 weeks. In the second arm, PSC 833 is administered PO four times a day for 3 days; paclitaxel is administered by continuous infusion over 3 hours on day 2. Courses repeat every 3 weeks.

PROJECTED ACCRUAL: Approximately 70 patients will be accrued per year in this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Metastatic breast cancer within 2 years of an adjuvant anthracycline based chemotherapy for advanced disease, or failure of one prior anthracycline based chemotherapeutic regimen for advanced breast cancer Exception: When anthracyclines are contraindicated, metastatic disease within 2 years of any adjuvant cytotoxic regimen, or failure of one prior cytotoxic chemotherapeutic regimen for advanced breast cancer also qualifies Evaluable or measurable disease in at least one nonirradiated area No CNS metastases

PATIENT CHARACTERISTICS: Age: Not specified Performance status: SWOG 0-2 Life expectancy: Not specified Hematopoietic: Platelet count at least 100,000/mm3 Hemoglobin at least 8.0 g/dL Absolute neutrophil count at least 1500/mm3 Hepatic: Total serum bilirubin no greater than 1.5 mg/dL No history of chronic active hepatitis or cirrhosis SGOT and/or SGPT no greater than 2 times the upper limit of normal Renal: Serum creatinine no greater than 2.0 mg/dL Other: Not HIV positive Not pregnant or nursing Effective contraceptive required of fertile patients No uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or bowel obstruction No history of a second malignancy with the exception of non-melanoma skin cancer or carcinoma in situ of the cervix No known hypersensitivity to ingredients of the study medication or cyclosporine No neurologic problems requiring treatment No treatment with drugs within 48 hours that are known to interact with cyclosporine

PRIOR CONCURRENT THERAPY: At least 4 weeks since any investigational therapy Biologic therapy: No concurrent antibiotics, e.g. clarithromycin, erythromycin, nafcillin, rifampin, itraconazole, ketoconazole, or fluconazole (no greater than 200 mg/day allowed) Chemotherapy: No prior paclitaxel At least 6 weeks since nitrosoureas At least 4 weeks since other myelosuppressive chemotherapy Endocrine therapy: At least 2 weeks since hormone therapy No concurrent danazol Radiotherapy: At least 3 weeks since radiation therapy Surgery: Must be recovered from previous surgery Other: No concurrent calcium channel blockers, e.g. diltiazem, nicardipine, and verapamil No concurrent anticonvulsants, e.g. carbamazepine, phenobarbital, and phenytoin No concurrent bromocriptine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 1996-06; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James H. Doroshow, MD, Study Chair — City of Hope Comprehensive Cancer Center
Locations (4):
- United States (3):
  - Beckman Research Institute, City of Hope, Duarte, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California
- Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario, Canada